CLINICAL TRIAL: NCT02941640
Title: Influence of the Different Ways of Appendix Stump Closure on Patient Outcome in Laparoscopic Appendectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Clinical Center Tuzla (Other)
Responsible Party: Principal Investigator, Samir Delibegovic, MD, Ph.D, Professor of surgery, Head of colorectal department, University Clinical Center Tuzla
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 04-09/2-12/16
Record Dates: First submitted 2016-10-12; First posted 2016-10-21 (Estimated); Results first posted 2017-06-14 (Actual); Last update posted 2017-06-14 (Actual); Status verified 2017-06

CONDITIONS: Appendicitis
Keywords: Laparoscopic appendectomy; Endoloop; Stapler; Hem-o-lok clip; DS clip
MeSH Terms: conditions — Appendicitis | interventions — Surgical Staplers

STUDY DESIGN:
Who Masked: Participant
Masking Description: The study included 120 patients randomly divided into four groups with 30 patients in each. The study was not blinded. The nurse designated for participation in this study allocated the patients randomly into four groups by selecting a sealed opaque envelope from a box and opening it in the operating theatre. A card inside the envelope contained name of the treatment. All the envelopes were prepared in advance in a ratio of 1:4, shuffled well, and placed in the box by the same nurse.
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Laparoscopic appendectomy. E group. (Experimental): The securing the base of appendix by Endo-loop.
  Interventions: Procedure: E group; Device: Endoloop
- Laparoscopic appendectomy. S group. (Experimental): The securing the base of appendix by stapler.
  Interventions: Procedure: S group; Device: Stapler
- Laparoscopic appendectomy. H group. (Experimental): The securing the base of appendix by Hem-o-lok clip.
  Interventions: Procedure: H group; Device: Hem-o-lok clip
- Laparoscopic appendectomy. DS group. (Experimental): The securing the base of appendix by DS clip.
  Interventions: Procedure: DS group; Device: DS clip

INTERVENTIONS:
Procedure: E group — The securing the base of appendix by endoloop.
  Other Names: Endoloop
  Arms: Laparoscopic appendectomy. E group.
Procedure: S group — The securing the base of appendix by Stapler.
  Other Names: Stapler
  Arms: Laparoscopic appendectomy. S group.
Procedure: H group — The securing the base of appendix by Hem-o-lok clip.
  Other Names: Hem-o-lok clip
  Arms: Laparoscopic appendectomy. H group.
Procedure: DS group — The securing the base of appendix by DS clip.
  Other Names: DS clip
  Arms: Laparoscopic appendectomy. DS group.
Device: Endoloop
  Arms: Laparoscopic appendectomy. E group.
Device: Stapler
  Arms: Laparoscopic appendectomy. S group.
Device: Hem-o-lok clip
  Arms: Laparoscopic appendectomy. H group.
Device: DS clip
  Arms: Laparoscopic appendectomy. DS group.

SUMMARY:
During laparoscopic appendectomy, the base of the appendix is usually secured by an endoloop ligature or the stapler. Non-absorbable plastic hem-o-lok clip was shown as an alternative technique with which laparoscopic appendectomy was done faster and cheaper than the standard techniques. However, biocompatibility of different materials udes in securing the base of appendix is different. It was observed that stapler's clips made by titanium caused the mildest inflammatory reaction and creation of adhesions. Disadvantages of stapler's are their high price.

Titanium clips made for the use in laparoscopic appendectomy are safe and effective option in securing the appendicular stump in laparoscopic appendectomy. They have potential advantages over stapler, because they have the same bio compatibility, and their price is lower.

DETAILED DESCRIPTION:
Prospective study was conducted in the period from 02. October 2016 to 30. December 2016. The patients were randomly divided into four groups; in the first group, the base of the appendix was secured using one endoloop ligature, in the second group using the 45-mm stapler, in third group using only one non-absorbable Hem-o-lok clip and in fourth group using titanium DS clip.

Patients were assessed for eligibility at the emergency station by the surgeon on-call once the diagnosis of acute appendicitis was established. A dedicated study nurse assigned randomly to Endoloop (E group) or Stapler (S group), or Hem-o-lock (H group), or DS clip (DS group) by picking out of a box and opening a sealed opaque randomization envelope in operating theatre. The details of the allocated treatments (''E'' or ''S'', or (''H'' or (''Ds'' ) were given on cards contained in sealed opaque envelopes. All sealed opaque envelopes were previously prepared with a 1 : 1 ratio, well shuffled, and put into a box by the dedicated study nurse. No blinding was performed.

Data collected included age, gender, surgery time, time of hem-o-lok clip application, hospital stay, costs associated with these and intra- and post-operative complications.

Technique

The patient was placed in supine position, combined with Trendelenburg position and left lateral position (10º - 15º, incline towards the surgeon). The surgeon used the French position (between legs of patient) and an assistant stood on the left side, and monitor was on the right side of the patient. The bladder was decompressed with the Foley catheter to avoid an injury during insertion of the supra-pubic ports. Pneumoperitoneum was established with the Veress needle through the umbilicus and then an endoscope was introduced. Under direct vision, one 12 mm trocar was inserted in suprapubic region, a little to the left, and 5 mm trocar in the right lower quadrant, to the level of the first 12 mm port, in order to acquire triangulation. After that the abdominal cavity was inspected.

When the decision was made to perform appendectomy, mesoappendix was mobilized and dissected using an harmonic scalpel (Ethicon, Endosurgery, Cincinnati, OH). In the first group, the base of the appendix was secured using one endoloop, and on the distal part which would be removed, another endoloop was used. In the second group, the appendix was secured by a 45 mm stapler (thick charge) (Ethicon, Endosurgery, Cincinnati, OH). In the third group, one hem-o-lok clip, size XL (Hem-o-lock, Weck Closure Systems, Research Triangle Park, NC, USA) was placed on the base the appendix by a special applier for the hem-o-lok clip, and on the distal part which would be removed, another clip was used. In the fourth group, one titanium DS clip (Aesculap AG, Tuttlingen, Germany) was placed on the base of appendix by endoscopic clip applier (12 mm) and on the distal part which would be removed, another DS clip was used.

ELIGIBILITY:
Inclusion Criteria:

* Patient with accute appendicits

Exclusion Criteria:

* Patient younger than 18 years

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2016-10-02 (Actual); Primary Completion 2016-12-30 (Actual); Study Completion 2017-01-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Enver Zerem, MD, PhD, Study Chair — University Clinical Center Tuzla
Locations (1):
- University Clinical Center Tuzla, Tuzla, Bosnia and Herzegovina

IPD SHARING:
Plan to Share IPD: No
We have no plan to share IPD.

RESULTS

PARTICIPANT FLOW:
Groups:
- Laparoscopic Appendectomy. Endoloop.: Laparoscopic appendectomy. The securing the base of appendix by endo-loop.
  Laparoscopic appendectomy: The securing the base of appendix by endoloop.
  Endoloop
- Laparoscopic Appendectomy. Stapler: Laparoscopic appendectomy. The securing the base of appendix by stapler.
  Laparoscopic appendectomy: The securing the base of appendix by Stapler.
  Stapler
- Laparoscopic Appendectomy. Hem-o-lok Clip: Laparoscopic appendectomy. The securing the base of appendix by Hem-o-lok clip.
  Laparoscopic appendectomy: The securing the base of appendix by Hem-o-lok clip.
  Hem-o-lok clip
- Laparoscopic Appendectomy. DS Clip: Laparoscopic appendectomy.The securing the base of appendix by DS clip.
  Laparoscopic appendectomy: The securing the base of appendix by DS clip.
  DS clip
Period: Overall Study
Arm/Group | Laparoscopic Appendectomy. Endoloop. | Laparoscopic Appendectomy. Stapler | Laparoscopic Appendectomy. Hem-o-lok Clip | Laparoscopic Appendectomy. DS Clip
Started | 30 | 30 | 30 | 30
Completed | 30 | 30 | 30 | 30
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Sex baseline measure
Groups:
- Total: Total of all reporting groups
Arm/Group | Laparoscopic Appendectomy. Endoloop. | Laparoscopic Appendectomy. Stapler | Laparoscopic Appendectomy. Hem-o-lok Clip | Laparoscopic Appendectomy. DS Clip | Total
Number analyzed (Participants) | 30 | 30 | 30 | 30 | 120
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.17 (13.45) | 30.93 (12.34) | 32.63 (13.97) | 29.53 (14.65) | 31.07 (13.50)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 15 | 17 | 13 | 61
  Male | 14 | 15 | 13 | 17 | 59

OUTCOME MEASURES:

1. Primary Outcome: Overall Morbidity
Description: Overall morbidity following the securing of the base of the appendix, defined as any adverse event occurring from the time of securing the base of the appendix until the 30th day.
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Laparoscopic Appendectomy. Endoloop. | Laparoscopic Appendectomy. Stapler | Laparoscopic Appendectomy. Hem-o-lok Clip | Laparoscopic Appendectomy. DS Clip
Number analyzed (Participants) | 30 | 30 | 30 | 30
Participants | 0 | 0 | 0 | 0

2. Secondary Outcome: Intra-perative Complications
Description: Complications that appear during operative procedure
Time Frame: 120 min.
Measure: Count of Participants; unit: Participants
Arm/Group | Laparoscopic Appendectomy. Endoloop. | Laparoscopic Appendectomy. Stapler | Laparoscopic Appendectomy. Hem-o-lok Clip | Laparoscopic Appendectomy. DS Clip
Number analyzed (Participants) | 30 | 30 | 30 | 30
Participants | 0 | 0 | 0 | 0

3. Secondary Outcome: Postoperative Complications
Description: Complications that appear after operative procedure
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Laparoscopic Appendectomy. Endoloop. | Laparoscopic Appendectomy. Stapler | Laparoscopic Appendectomy. Hem-o-lok Clip | Laparoscopic Appendectomy. DS Clip
Number analyzed (Participants) | 30 | 30 | 30 | 30
Participants | 0 | 0 | 0 | 0

4. Secondary Outcome: Operative Time
Description: Time of operative procedure
Time Frame: 120 min.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Laparoscopic Appendectomy. Endoloop. | Laparoscopic Appendectomy. Stapler | Laparoscopic Appendectomy. Hem-o-lok Clip | Laparoscopic Appendectomy. DS Clip
Number analyzed (Participants) | 30 | 30 | 30 | 30
minutes | 46.0 (7.07) | 39.37 (7.2) | 42.83 (6.52) | 47.47 (6.2)
Statistical Analysis 1: Comparison: Laparoscopic Appendectomy. Endoloop. vs Laparoscopic Appendectomy. Stapler vs Laparoscopic Appendectomy. Hem-o-lok Clip vs Laparoscopic Appendectomy. DS Clip; Test type: Other — Anova; p < 0.0001, ANOVA — Significant when P<0.05
Statistical Analysis 2: Comparison: Laparoscopic Appendectomy. Endoloop. vs Laparoscopic Appendectomy. Stapler; Post hoc analysis was done by Tukey test; Test type: Other; p = 0.001, Tukey post hoc test — Significant when P<0.05
Statistical Analysis 3: Comparison: Laparoscopic Appendectomy. Stapler vs Laparoscopic Appendectomy. DS Clip; Test type: Other — Tukey post hoc test; p < 0.0001, Tukey post hoc test — Significant when P<0.05
Statistical Analysis 4: Comparison: Laparoscopic Appendectomy. Hem-o-lok Clip vs Laparoscopic Appendectomy. DS Clip; Test type: Other; p = 0.044, Tukey post hoc test — Significant when P<0.05
Statistical Analysis 5: Comparison: Laparoscopic Appendectomy. Endoloop. vs Laparoscopic Appendectomy. Hem-o-lok Clip; Test type: Other; p < 0.272, Tukey post hoc test — Significant when P<0.05
Statistical Analysis 6: Comparison: Laparoscopic Appendectomy. Endoloop. vs Laparoscopic Appendectomy. DS Clip; Test type: Other; p = 0.835, Tukey post hoc test — Significant when P<0.05
Statistical Analysis 7: Comparison: Laparoscopic Appendectomy. Stapler vs Laparoscopic Appendectomy. Hem-o-lok Clip; Test type: Other; p = 0.199, Tukey post hoc test — Significant when P<0.05

5. Secondary Outcome: Time of Application
Description: Time of application of endoloop, stapler, Hem-o-lok and DS clip measured from introducing of instruments to cutting the base of appendix
Time Frame: 120 min
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Laparoscopic Appendectomy. Endoloop. | Laparoscopic Appendectomy. Stapler | Laparoscopic Appendectomy. Hem-o-lok Clip | Laparoscopic Appendectomy. DS Clip
Number analyzed (Participants) | 30 | 30 | 30 | 30
seconds | 195.50 (62.13) | 19.87 (4.64) | 63.90 (10.31) | 63.77 (27.80)
Statistical Analysis 1: Comparison: Laparoscopic Appendectomy. Endoloop. vs Laparoscopic Appendectomy. Stapler vs Laparoscopic Appendectomy. Hem-o-lok Clip vs Laparoscopic Appendectomy. DS Clip; Test type: Other — Anova; p < 0.0001, ANOVA — Significant when P<0.05
Statistical Analysis 2: Comparison: Laparoscopic Appendectomy. Endoloop. vs Laparoscopic Appendectomy. Stapler; Test type: Other; p < 0.0001, Tukey post hoc test — Significant when P<0.05
Statistical Analysis 3: Comparison: Laparoscopic Appendectomy. Endoloop. vs Laparoscopic Appendectomy. Hem-o-lok Clip; Test type: Other; p < 0.0001, Tukey post hoc test — Significant when P<0.05
Statistical Analysis 4: Comparison: Laparoscopic Appendectomy. Endoloop. vs Laparoscopic Appendectomy. DS Clip; Test type: Other; p < 0.0001, Tukey post hoc test — Significant when P<0.05
Statistical Analysis 5: Comparison: Laparoscopic Appendectomy. Stapler vs Laparoscopic Appendectomy. Hem-o-lok Clip; Test type: Other; p < 0.0001, Tukey post hoc test
Statistical Analysis 6: Comparison: Laparoscopic Appendectomy. Stapler vs Laparoscopic Appendectomy. DS Clip; Test type: Other; p < 0.0001, Tukey post hoc test — Significant when P<0.05
Statistical Analysis 7: Comparison: Laparoscopic Appendectomy. Hem-o-lok Clip vs Laparoscopic Appendectomy. DS Clip; Test type: Other; p = 1.00, Tukey post hoc test — Significant when P<0.05

6. Secondary Outcome: Hospital Stay
Description: Length of hospitalization
Time Frame: 30 days
Measure: Median (Standard Deviation); unit: days
Arm/Group | Laparoscopic Appendectomy. Endoloop. | Laparoscopic Appendectomy. Stapler | Laparoscopic Appendectomy. Hem-o-lok Clip | Laparoscopic Appendectomy. DS Clip
Number analyzed (Participants) | 30 | 30 | 30 | 30
days | 2.17 (0.70) | 2.20 (0.71) | 2.23 (0.78) | 2.37 (0.72)

ADVERSE EVENTS:
Time Frame: Adverse event information was collected on post-operative days 1, 2, 7, 14, and 30th day.
Description: A standard questionnaire and regular investigator assessment was collected from all participants in the study to assess/monitor adverse events.
Arm/Group | Laparoscopic Appendectomy. Endoloop. | Laparoscopic Appendectomy. Stapler | Laparoscopic Appendectomy. Hem-o-lok Clip | Laparoscopic Appendectomy. DS Clip
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30 | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30 | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30 | 0/30 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No